CLINICAL TRIAL: NCT05668364
Title: Outdoor Cold Air Exposure Versus Room Temperature for Croup Symptoms in Pediatric Emergency Departments: a Randomized Controlled Trial
Brief Title: Impact of Cold Air Exposure on Croup Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pediatric Clinical Research Platform (Other)
Responsible Party: Principal Investigator, Johan Siebert, MD, Deputy Head of the Pediatric Emergency Department, Pediatric Clinical Research Platform
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-00845
Record Dates: First submitted 2022-12-12; First posted 2022-12-29 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Croup
Keywords: Croup; Laryngitis; Laryngotracheitis; Laryngotracheobronchitis; Pediatrics; Children; Infant; Cold air
MeSH Terms: conditions — Croup; Laryngitis

STUDY DESIGN:
Intervention Model Description: Open-label randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposition group (Experimental): Outdoor cold air exposure (<10°C or <50°F) for 30 minutes. On completion of the intervention, participants remained under observation at indoor ambient air from 30 minutes to 60 minutes from the intervention.
  Interventions: Other: Outdoor cold air exposure
- Control group (No Intervention): Indoor ambient air exposure (24-25°C or 75-77°C). Participants remained under observation at indoor ambient until 60 minutes from triage.

INTERVENTIONS:
Other: Outdoor cold air exposure — Exposure to outdoor cold air (<10°C or <50°F, intervention group) for 30 minutes. On completion of the intervention, participants remained under observation at indoor ambient air from 30 minutes to 60 minutes from the intervention.
  Arms: Exposition group

SUMMARY:
The goal of the present randomised controlled clinical trial is to compare the efficacy of a 30-minute exposition to cold, atmospheric, outdoor air on the severity of croup symptoms with exposition to indoor room air in children with mild to moderate croup receiving a single dose of dexamethasone during winter croup outbreaks.

DETAILED DESCRIPTION:
Croup is a viral laryngitis that represents the most common cause of acute upper airway obstruction in children. It is therefore a frequent reason for emergency department visits. The benefit of dexamethasone on croup symptoms is well established with an onset of action of at least 30 minutes. Various non-pharmacological measures, including exposition to cold air, are also thought to be effective in reducing the severity of symptoms, although this has not been demonstrated yet in the current scientific literature. The aim of the present study is to evaluate the efficacy of exposition to cold air on the symptoms of croup in children.

The investigators designed a prospective, open-label, single centre randomised controlled trial to evaluate the effect of exposition to cold air on the symptoms of croup in children.

The study was performed during autumn and winter croup outbreaks when outdoor air temperature was <10°C (<50°F). Participants were infants and children aged 3 months to 10 years presenting to the pediatric emergency department of our institution. Inclusion criteria were patients presenting with mild to moderate croup symptoms with Westley croup scores > or=2 (to permit a clinically relevant reduction in the Westley croup score of at least 2 points from baseline at 30 minutes), diagnosed by a triage nurse and confirmed by a senior attending pediatric emergency physician. Exclusion criteria were history or physical examination suggesting any other diagnosis, severe croup requiring immediate nebulised epinephrine, chronic respiratory disease (except asthma), underlying airway abnormalities, immunodeficiency; and contraindication to steroids. According to the recommended standards of care, all children with croup were administered a standard 0·6 mg/kg/dose oral dexamethasone at triage.

Participants were randomly allocated either to the outdoor cold air exposition group or to the indoor group allocation using a single, constant 1:1 allocation ratio. Demographic data, previous exposition to cold air before presentation at pediatric emergency department, as well as vital signs and Westley croup score on arrival, and after 30 and 60 minutes, were recorded. Parents were reached by phone 7 days after the initial visit to assess the child's clinical outcome and the final diagnosis, as well as the need for further consultation or hospitalization in the meantime.

ELIGIBILITY:
Inclusion Criteria:

- children from 3 months to 10 years with clinical signs of croup and Westley croup score > or =2

Exclusion Criteria:

* Need for close monitoring
* Need for nebulized epinephrine
* History or physical examination suggesting any other diagnosis
* Chronic respiratory disease (except asthma)
* Underlying airway abnormalities
* Immunodeficiency
* Contraindication to steroids

Ages: 3 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Westley croup score at 30 minutes | at 30 minutes
  The primary outcome is the proportion of patients showing an decrease of at least 2 points in their Westley croup score at 30 minutes from triage.
  The 5-item Westley croup score uses a 17 points ordinal scale to assess level of consciousness (5 points), cyanosis (5 points), stridor (2 points), air entry (2 points), and chest wall retractions (3 points). Mild croup is defined as a WCS < or = 2, moderate 3-5, severe 6-11, and impending respiratory failure or >12.

SECONDARY OUTCOMES:
Westley croup score at 60 minutes | at 60 minutes
  The secondary outcome is the proportion of patients showing an decrease of at least 2 points in their Westley croup score at 60 minutes from triage.
  The 5-item Westley croup score uses a 17 points ordinal scale to assess level of consciousness (5 points), cyanosis (5 points), stridor (2 points), air entry (2 points), and chest wall retractions (3 points). Mild croup is defined as a WCS < or = 2, moderate 3-5, severe 6-11, and impending respiratory failure or >12.
Pulse oxymetry | at 0 min, at 30 and at 60 minutes from enrolment at triage
  Pulse oxymetry in %
Respiratory rate | at 0 min, at 30 and at 60 minutes from enrolment at triage
  Respiratory rate in breaths/min
Heart rate | at 0 min, at 30 and at 60 minutes from enrolment at triage
  Heart rate in beats/min
Telephone Outpatient derived score | at the time of leaving home for the pediatric emergency department visit; at 0 min on pediatric emergency department arrival (i.e., at triage); at day 7 from the initial visit
  Anamnestic scoring tool to estimate croup severity, derived from the original Telephone Out Patient score
Hospitalisation rate | Within 7 days from the initial visit
  Rate of hospital admission for croup
Adverse events | at 30 minutes from enrolment at triage
  Parental or patient perception of adverse events related to exposure to outdoor cold air.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Siebert, MD, Principal Investigator — University Hospitals of Geneva

IPD SHARING:
Plan to Share IPD: Yes
Deidentified Individual Participant Data will be available from the corresponding author upon reasonable request, recognizing that these data will only provide results for the current trial and not for future trials. Only deidentified/anonymized data will be shared.
Supporting Information: Study Protocol
Time Frame: 6 month to 5 years after publication of results.
Access Criteria: Data will be made available from the corresponding author upon approval of a proposal and after a signed data access agreement.
  Deidentified participant data will be made available to qualified external researchers who will use them according to their Institutional Review Board.
  Data will be made available for a specified research purpose. The request proposal should include participation of a statistician.

REFERENCES:
- [Background] Gates A, Gates M, Vandermeer B, Johnson C, Hartling L, Johnson DW, Klassen TP. Glucocorticoids for croup in children. Cochrane Database Syst Rev. 2018 Aug 22;8(8):CD001955. doi: 10.1002/14651858.CD001955.pub4. PMID 30133690
- [Result] Hanna J, Brauer PR, Morse E, Berson E, Mehra S. Epidemiological analysis of croup in the emergency department using two national datasets. Int J Pediatr Otorhinolaryngol. 2019 Nov;126:109641. doi: 10.1016/j.ijporl.2019.109641. Epub 2019 Aug 13. PMID 31442871
- [Result] Johnson DW. Croup. BMJ Clin Evid. 2014 Sep 29;2014:0321. PMID 25263284
- [Result] Moore M, Little P. Humidified air inhalation for treating croup. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD002870. doi: 10.1002/14651858.CD002870.pub2. PMID 16855994
- [Result] Bjornson CL, Williamson J, Johnson DW. Telephone Out Patient Score: The Derivation and Validation of a Telephone Follow-up Assessment Tool for Use in Clinical Research in Children With Croup. Pediatr Emerg Care. 2016 May;32(5):290-7. doi: 10.1097/PEC.0000000000000796. PMID 27139290
- [Derived] Siebert JN, Salomon C, Taddeo I, Gervaix A, Combescure C, Lacroix L. Outdoor Cold Air Versus Room Temperature Exposure for Croup Symptoms: A Randomized Controlled Trial. Pediatrics. 2023 Sep 1;152(3):e2023061365. doi: 10.1542/peds.2023-061365. PMID 37525974